CLINICAL TRIAL: NCT07034326
Title: Observation on the Clinical Efficacy of Electroacupuncture Combined With Immune Checkpoint Inhibitors as Adjuvant Therapy After Surgery for Early-stage Non-small Cell Lung Cancer
Brief Title: Electroacupuncture Combined With Immune Checkpoint Inhibitors as Adjuvant Therapy After Surgery for Early-stage Non-small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kong Fanming (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Sponsor-Investigator, Kong Fanming, Director of Oncology Department, First Teaching Hospital of Tianjin University of Traditional Chinese Medicine
Organization: First Teaching Hospital of Tianjin University of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TYLL2024[Z]082
Record Dates: First submitted 2025-06-15; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Non-Small Cell Lung Cancer; Electroacupuncture; Immune Checkpoint Inhibitors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Electroacupuncture combined with immunotherapy (Experimental)
  Interventions: Other: Electroacupuncture combined with immunotherapy
- Zilongjin tablet combined with immunotherapy (Experimental)
  Interventions: Drug: Zilongjin tablet combined with immunotherapy
- Immunotherapy (Active Comparator)
  Interventions: Drug: Immunotherapy

INTERVENTIONS:
Other: Electroacupuncture combined with immunotherapy — Connect the electroacupuncture therapy instrument, select the density wave 2 Hz/100 Hz, the current intensity should be tolerated by the patient, leave the needle for 20 min.Immunotherapy including but not limited to pabolizumab and attilizumab were repeated every 21 days for treatment weeks.The period is 1 year, and maintenance treatment can be carried out in accordance with the drug instructions and guidelines.
  Arms: Electroacupuncture combined with immunotherapy
Drug: Zilongjin tablet combined with immunotherapy — Take Zilongjin tablets orally, 4 tablets each time, 3 times a day.Immunotherapy including but not limited to pabolizumab and attilizumab were repeated every 21 days for treatment weeks.The period is 1 year, and maintenance treatment can be carried out in accordance with the drug instructions and guidelines.
  Arms: Zilongjin tablet combined with immunotherapy
Drug: Immunotherapy — Immunotherapy including but not limited to pabolizumab and attilizumab were repeated every 21 days for treatment weeks.The period is 1 year, and maintenance treatment can be carried out in accordance with the drug instructions and guidelines.
  Arms: Immunotherapy

SUMMARY:
Postoperative immunoadjuvant therapy has been proven to significantly reduce the risk of recurrence after resectable NSCLC, and has become a new standard of postoperative adjuvant therapy for stage II-III NSCLC. Immunotherapy faces challenges such as immune resistance, heterogeneity of biomarker expression, and limitation of immune-suitable population. How to reduce the rate of recurrence and metastasis after surgery, enhance the therapeutic effect of immunotherapy, and then prolong the survival period and improve the quality of life, has become an urgent problem facing the current clinical. Based on the standards of evidence-based medicine, this study for the first time carried out a large sample, multi-center, randomized parallel controlled clinical study to obtain high-quality clinical evidence of the effectiveness and safety of electro-acupuncture and Zilongjin tablet synergic treatment, and formed a standard treatment plan of traditional Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

* (1) Non-tumor patients with stage Ⅱ, ⅢA, ⅢB (N2) non-small cell lung cancer diagnosed by pathology or cytology after surgery; (2) driver mutations negative patients; (3) Postoperative adjuvant chemotherapy was received for 1 to 4 cycles;(4)conforms to two qi syndrome of traditional Chinese medicine syndrome differentiation diagnosis of patients; (5) aged 18 to 80 years old; (6) expected lifetime > 6 months; (7) ECOG 0 to 2 points; (8) patients willing to accept this solution treatment, adherence to the good.

Exclusion Criteria:

* (1) Patients with other malignant tumors in the past or at the same time within 5 years; (2) has a serious heart, liver and kidney damage, or other serious complications; (3) the R1, R2, need after resection, postoperative adjuvant radiotherapy patients; (4) with mental disorders; (5) has a variety of drug allergy, allergic constitution; (6) in pregnancy or lactation women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease free survival(DFS) | 2year
  Time from random start to first recurrence or death.

SECONDARY OUTCOMES:
DFS | 3year
  Time from random start to first recurrence or death.
Overall survival | 3,5year
EORTC QLQ-C30 Scale | 0,2,3,6 month
  EORTC QLQ-C30 Scale
Immune function | 0,3 month
  T lymphocyte subsets, NK cells
Lung cancer TCM syndrome score | 0,2,3,6 month

CONTACTS AND LOCATIONS:
Locations (1):
- First Teaching Hospital of Tianjin University of Traditional Chinese Medicine, Tianjin, China

IPD SHARING:
Plan to Share IPD: No